CLINICAL TRIAL: NCT01536249
Title: An Open-Label Study to Assess the Effect of Cimetidine on the Pharmacokinetics of Dexpramipexole (BIIB050) in Healthy Volunteers
Brief Title: Dexpramipexole and Cimetidine Drug Drug Interaction (DDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 223HV104
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Dexpramipexole; Cimetidine

ARMS (2):
- Dexpramipexole single dose & 12 Doses Cimetidine (Experimental): 300 mg Dexpramipexole Oral Dose (to be taken in conjunction with multiple doses of Cimetidine at 400 mg per dose)
  Interventions: Drug: Cimetidine plus Dexpramipexole
- Dexpramipexole single Dose (Experimental): 300 mg Dexpramipexole Oral Dose
  Interventions: Drug: Dexpramipexole

INTERVENTIONS:
Drug: Dexpramipexole — Single Oral Dose
  Arms: Dexpramipexole single Dose
Drug: Cimetidine plus Dexpramipexole — Multiple Oral Doses
  Arms: Dexpramipexole single dose & 12 Doses Cimetidine

SUMMARY:
This study will assess the effect of cimetidine on the pharmacokinetics (PK) of dexpramipexole in healthy volunteer and evaluate the safety and tolerability of dexpramipexole when given with or without cimetidine. Additionally, this study will explore the influence of genetic variation on the PK of dexpramipexole when given with or without cimetidine.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, two-period, crossover study in approximately 14 healthy subjects. The goals of this study are as follows:

To assess the effect of cimetidine on the pharmacokinetics (PK) of dexpramipexole in healthy volunteers.

To evaluate the safety and tolerability of dexpramipexole when given with or without cimetidine.

To explore the influence of genetic variation on the PK of dexpramipexole when given with or without cimetidine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the Investigator, are healthy as determined by medical history, physical examination, and 12 lead ECG
* Adult males/females aged 18 to 55 years inclusive
* Male and female subjects of childbearing potential must practice effective contraception during the study and up to 90 days after their last dose.

Exclusion Criteria:

* History of malignant disease, including solid tumors and hematologic malignancies.
* History of clinically significant endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major diseases, as determined by the Investigator.
* Treatment with prescription medication and/or over-the-counter products and herbal-containing and/or alternative health preparations and procedures.
* Surgery within 90 days prior to check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determination of the effect of cimetidine on the PK of dexpramipexole parameters including: AUC: Area under the plasma-concentration time curve over a specified time period; Cmax: Maximum observed plasma concentration and CLr: renal clearance | pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, and 72 hours after dexpramipexole administration in each dosing period.

SECONDARY OUTCOMES:
PK parameters of dexpramipexole including, but not limited to, half-life when given with or without cimetidine | pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, and 72 hours after dexpramipexole administration in each dosing period.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States